CLINICAL TRIAL: NCT04846582
Title: A New Method for Evaluating Endometriosis Using MRI: A Study on the MEDL Score
Brief Title: An Observational Study of Patients With Endometriosis to Evaluate the Usefulness of the MEDL Score, a New Method for Evaluating Endometriosis Using MRI
Status: Completed | Type: Observational
Sponsor: Chugai Pharmaceutical (Industry)
Collaborators: Clinica Medicina da Mulher (Unknown)
Responsible Party: Sponsor
Other Study IDs: AMY007BR
Record Dates: First submitted 2021-02-18; First posted 2021-04-15 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other

SUMMARY:
The purpose of this study is to confirm the reproducibility that the MEDL score can be evaluated by Magnetic Resonance Imaging (MRI) in the similar way as laparoscopy, the gold standard for the evaluation of the disease state of endometriosis, in order to establish the MEDL score, a new evaluation index for endometriosis using MRI. Approximately 70-90 patients with endometriosis diagnosed by imaging and who are candidates for fertility-preserving surgery will be recruited retrospectively or prospectively, and the disease status of endometriosis will be evaluated using preoperative MR images, laparoscopic surgery videos, etc. The relationship between the condition and clinical symptoms, such as pain, is also considered.

ELIGIBILITY:
Inclusion Criteria:

* Patients who consent to use their data in this study
* Patients with endometriosis diagnosed by transvaginal ultrasound (TVUS) and/or MRI
* Patients undergoing fertility-preserving surgery
* Patients with pain due to endometriosis
* Patients with endometriotic lesions other than ovarian cysts confirmed by MRI (concomitant ovarian cysts can be recruited)
* Patients with the following patient clinical information (TVUS is not mandatory when archived data is used)

Patient clinical information: Preoperative MR images, videos of laparoscopic surgery, pathological evaluation of endometriosis, videos of preoperative TVUS, pain information related to endometriosis, information about infertility before surgery, information on QOL, information on postoperative recurrence, information on surgical difficulty, operating time, length of hospital stay for surgical operation, age, history of treatment (drugs, surgery), anamnesis and complication, history of endometriosis, age at menarche, menstrual cycle, date of surgery, date of MR image acquisition, operative procedure and history of pregnancy and childbirth.

Exclusion Criteria:

* Patients who had surgery for endometriosis prior to the surgery included in this study
* Patients deemed inappropriate by the principal investigator
* Patients who obtained their voluntary consent but later withdrew their consent

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with endometriosis diagnosed by imaging and who are candidates for fertility-preserving surgery
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-01-10 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Correlation of MEDL score assessed by MRI and laparoscopy | at the time of surgery
  Correlation coefficient of total MEDL score assessed by preoperative MRI and laparoscopy

SECONDARY OUTCOMES:
Association of MRI findings by MEDL score with pain | preoperative
  Correlation coefficient between preoperative pain Visual Analog Scale (VAS) score and total MEDL score
Association of MRI findings by MEDL score with infertility | preoperative
  Relationship between presence or absence of infertility and total MEDL score
Association of MRI findings by MEDL score with SF-36 | preoperative
  Relationship between responses to the SF-36 questionnaire and total MEDL score
Association of MRI findings by MEDL score with Endometriosis Health Profile Questionnaire-30 (EHP-30) | preoperative
  Relationship between responses to the EHP-30 questionnaire and total MEDL score
Association of MRI findings by MEDL score with postoperative recurrence | from surgery to obtaining informed consent, assessed up to 3 years (for retrospective data collection)
  Relationship between presence or absence of postoperative recurrence
Association of MRI findings by MEDL score with Ultrasound-based Endometriosis Staging System (UBESS) | preoperative
  Relationship between stage of UBESS and total MEDL score
Association of MRI findings by MEDL score with operating time | at the time of surgery
  Relationship between hospital stay and total MEDL score
Association of MRI findings by MEDL score with hospital stay | at the time of surgery
  Relationship between hospital stay and total MEDL score
Agreement rate among evaluators using the MEDL score | at the time of preoperative MR imaging
  The agreement rate for each evaluation item of MEDL score when multiple evaluators evaluated
K coefficient among evaluators using the MEDL score | at the time of preoperative MR imaging
  K coefficient for each evaluation item of MEDL score when multiple evaluators evaluated
Concordance between laparoscopic findings and transvaginal ultrasound findings using the MEDL score | at the time of surgery
  Correlation coefficient of total MEDL score assessed by preoperative transvaginal ultrasound and laparoscopy
Association of MRI findings by MEDL score with rASRM score evaluated by laparoscopy | at the time of surgery
  Correlation coefficient of total MEDL score assessed by preoperative MRI and rASRM score assessed by laparoscopy
Association of MRI findings by MEDL score with ENZIAN classification evaluated by laparoscopy and MRI | at the time of surgery
  Association between total MEDL score assessed by preoperative MRI and ENZIAN classification assessed by laparoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor Chugai Pharmaceutical Co. Ltd, Study Director — clinical-trials@chugai-pharm.co.jp
Locations (1):
- Clinica Medicina da Mulher, São Sebastião, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform. For further details on Chugai's Data Sharing Policy and how to request access to related clinical study documents, see here (www.chugai-pharm.co.jp/english/profile/rd/ctds_request.html).